CLINICAL TRIAL: NCT05694923
Title: Effect of Sodium Glucose Cotransporter Inhibitors on Fatty Liver Disease Patients
Brief Title: Effect of Sodium Glucose Cotransporter Inhibitors Fatty Liver Disease Patients Fatigue Assessment
Acronym: Fatty liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa osman taha, Lecturer of internal medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Assiut 1989
Record Dates: First submitted 2023-01-09; First posted 2023-01-23 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Fatty Liver Disease
Keywords: Fatty Liver Nonalcoholic nondiabetic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Single center clinical randomized trial open labelled study patients of non diabetic non alcoholic fatty liver from outpatient clinic at assiut university will be randomized and recruited into arms Group A Will receive empaglifizon sodium glucose cotransporter in minimum dose 10 mg Group B Will be Instructed for diet control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- life style modification and diet control (No Intervention): 33 patient of non alcoholic fatty liver patients and non diabetic only receive life style modification and diet control
- empaglifizon 10 mg plus life style and diet control (Experimental): 22 patient of non alcoholic fatty liver patients and non diabetic Will receive empaglifizon in minimum dose 10 mg in addition to life style modification and diet control
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — non fatty liver non alcoholic patients Will receive empaglifizon sodium glucose cotransporter in minimum dose 10 mg
  Arms: empaglifizon 10 mg plus life style and diet control

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has become a major health problem worldwide with an increasing prevalence ranging from 13% in Africa to 42% in South-East Asia. The term NAFLD includes a variety of diseases, ranging from liver fat deposition in more than 5% of hepatocytes (steatosis-non-alcoholic fatty liver (NAFL)) to necroinflammation and fibrosis (non-alcoholic steatohepatitis (NASH)), which can progress into NASH-cirrhosis, and eventually to hepatocellular carcinoma 1 Lifestyle modifications remain the cornerstone of NAFLD treatment, even though various pharmaceutical interventions are currently under clinical trial. Among them, sodium-glucose co-transporter type-2 inhibitors (SGLT-2i) are emerging as promising agents. Processes regulated by SGLT-2i, such as endoplasmic reticulum (ER) and oxidative stress, low-grade inflammation, autophagy and apoptosis are all implicated in NAFLD pathogenesis 2

In non-DM patients, only a small single center study exists which studied 12 patients under dapagliflozin and 10 patients under teneligliptin, a DPP4 inhibitor, for a total of 12 weeks, showing that after this intervention period, serum transaminases were decreased in both groups, while in the dapagliflozin group, total body water and body fat decreased, leading to decreased total body weight.3

DETAILED DESCRIPTION:
Introduction :

Non-alcoholic fatty liver disease (NAFLD) has become a major health problem worldwide with an increasing prevalence ranging from 13% in Africa to 42% in South-East Asia. The term NAFLD includes a variety of diseases, ranging from liver fat deposition in more than 5% of hepatocytes (steatosis-non-alcoholic fatty liver (NAFLD)) to necroinflammation and fibrosis (non-alcoholic steatohepatitis (NASH)), which can progress into NASH-cirrhosis, and eventually to hepatocellular carcinoma 1 Lifestyle modifications remain the cornerstone of NAFLD treatment, even though various pharmaceutical interventions are currently under clinical trial. Among them, sodium-glucose co-transporter type-2 inhibitors (SGLT-2i) are emerging as promising agents. Processes regulated by SGLT-2i, such as endoplasmic reticulum (ER) and oxidative stress, low-grade inflammation, autophagy and apoptosis are all implicated in NAFLD pathogenesis 2

In non-DM patients, only a small single center study exists which studied 12 patients under dapagliflozin and 10 patients under teneligliptin, a DPP4 inhibitor, for a total of 12 weeks, showing that after this intervention period, serum transaminases were decreased in both groups, while in the dapagliflozin group, total body water and body fat decreased, leading to decreased total body weight.3

Aim of the study :

To evaluate efficacy of sodium glucose cotransporter inhibitors to improve outecomes among non diabetic non alcoholic fatty liver patients

Designs Single center clinical randomized trial open labelle patients of non diabetic non alcoholic fatty liver from outpatient clinic at assiut university will be randomized and recruited into arms Group A Will receive empaglifizon sodium glucose cotransporter in minimum dose 10 mg Group B Will be Instructed for diet control

All patients will be initially evaluated Full history medical history include Age .Sex Family history of DM ,HX OF HTN DRUG INTAKE history of ALCOHOL intake ..smoking Hx of fatigue Examination weight ,BMI ,waist circumference ,skin manifestation of insulin resistance

Investigation :

Liver enzymes (AlT …AST) Serology HCV Ab,HBsAg Fasting blood glucose ,2 hour blood glucoe HBA1C Lipid profile ,urine analysis TSH fatigue scal assessment ABDOMINAL US WILL BE DONE FOR ALL PATINTS Assesment of liver steatosis and fibrosis Fibroscan will be done initially for all cases

ELIGIBILITY:
Inclusion Criteria:

* non alcoholic fatty liver patients diagnosed at outpatient clinic of Assiut university

Exclusion Criteria:

- DM Patient Patient with viral hepatitis C,B Patient with hypothyroidism Patient with hepatotoxic drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy of sodium glucose cotransporter inhibitors to reduce hepatic steatosis and fibrosis among non diabetic non alcoholic fatty liver patients | 3 MONTHS
  assessment of fibrosis and steatosis by fiboscan as A CAP score that falls anywhere between 238 to 260 dB/m represents 11-33% fatty change in the liver. A CAP score that falls anywhere between 260 to 290 dB/m represents 34-66% fatty change in the liver. A CAP score that is 290 dB/m or higher represents over 67% fatty change in the liver

SECONDARY OUTCOMES:
fatigue assessment | 6 month
  fatigue follow up score more than 25 mild fatigue score range from 0 till 50 points

CONTACTS AND LOCATIONS:
Overall Officials: bahaa osman taha, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Asyut
  - Bahaa Osman, Asyut

REFERENCES:
- [Derived] Taha BO, Kobeisy MA, Abdelmohsen E, Abdelrhman T, Abokresha MM, Hassanein ZM, AbdEllah-Alawi MHM. Outcomes of empagliflozin in nondiabetic fatty liver patients: A randomized controlled trial. J Taibah Univ Med Sci. 2025 Aug 7;20(4):525-532. doi: 10.1016/j.jtumed.2025.07.008. eCollection 2025 Aug. PMID 40823521